CLINICAL TRIAL: NCT02494596
Title: A Phase Ib, Open-Label, Multicenter Study of the Safety and Pharmacokinetics of the Combination of RhuMab 2C4 (Omnitarg), a Recombinant Humanized Antibody to HER2, and Capecitabine (Xeloda) in Patients With Advanced Solid Tumors
Brief Title: A Phase Ib, Open-label, Multicenter Study of the Safety and PK of the Combination of rhuMAb2c4 (Omnitarg), a Recombinant Humanized Antibody to HER2, and Capecitabine (Xeloda) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17003
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Capecitabine; pertuzumab

ARMS (3):
- RhuMab 2C4 + Capecitabine 1000 mg/m^2 (Level 2) (Experimental): Participants will receive a single 1000-mg/m^2 dose of oral (PO) capecitabine on Day -7 for pretreatment assessment. Capecitabine will then be administered on Days 1 to 14 of each 3-week cycle at a dose of 1000 mg/m^2 twice daily, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 1050-mg IV infusion. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Capecitabine; Drug: RhuMab 2C4
- RhuMab 2C4 + Capecitabine 1250 mg/m^2 (Level 3) (Experimental): Participants will receive a single 1250-mg/m^2 dose of PO capecitabine on Day -7 for pretreatment assessment. Capecitabine will then be administered on Days 1 to 14 of each 3-week cycle at a dose of 1250 mg/m^2 twice daily, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 1050-mg IV infusion. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Capecitabine; Drug: RhuMab 2C4
- RhuMab 2C4 + Capecitabine 825 mg/m^2 (Level 1) (Experimental): Participants will receive a single 825-mg/m^2 dose of PO capecitabine on Day -7 for pretreatment assessment. Capecitabine will then be administered on Days 1 to 14 of each 3-week cycle at a dose of 825 mg/m^2 twice daily, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 1050-mg IV infusion. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Capecitabine; Drug: RhuMab 2C4

INTERVENTIONS:
Drug: Capecitabine — Participants will receive capecitabine on Days 1 to 14 of each 3-week cycle as 825, 1000, or 1250 mg/m^2 PO twice daily. Treatment may continue until disease progression, unacceptable toxicity, or consent withdrawal.
  Other Names: Xeloda
Drug: RhuMab 2C4 — Participants will receive rhuMab 2C4 on Day 1 of each 3-week cycle as 1050 mg via IV infusion. Treatment may continue until disease progression, unacceptable toxicity, or consent withdrawal.
  Other Names: Omnitarg

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of the combination of rhuMab 2C4(Perjeta) and capecitabine (Xeloda) in participants with advanced solid tumors that have progressed during or after standard therapy, or for which no standard therapy is available. Participants will be enrolled and evaluated for dose-limiting toxicities (DLTs) in escalating-dose cohorts in order to determine the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Easter Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 12 weeks
* Locally advanced or metastatic solid tumor with at least 1 measurable lesion, which has progressed during/after standard therapy
* Human epidermal growth factor receptor 2 (HER2)-negative among participants with breast cancer
* Negative pregnancy test or use of an adequate contraceptive method among women of childbearing potential
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Clinical evidence of central nervous system (CNS) metastases
* Prior chemotherapy, radiotherapy, or immunotherapy within 4 weeks, or hormone therapy within 2 weeks of study Day 1
* History of palmar plantar syndrome Grade 2 or worse, or any unresolved residual chemotherapy effects
* Prior HER2-active agents, continuous intravenous (IV) 5-fluorouracil, capecitabine, or other fluoropyrimidine
* Any investigational agent within 28 days of study start
* Prior cumulative doxorubicin dose greater than (>) 360 mg/m^2 or equivalent
* Significant cardiovascular disease
* Active/uncontrolled concurrent illness or infection-
* Major surgery or trauma within 4 weeks of study Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Barcelona, Spain
- Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were grouped into three cohorts and received either 825 mg, 1000 mg or 1250 mg capecitabine to determine the maximum tolerated dose.
Groups:
- Capecitabine 825 Plus (+) Pertuzumab 1050: Participants received a single dose of capecitabine 825 milligrams per square meter (mg/m^2) orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg intravenous (IV) infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
- Capecitabine 1000 + Pertuzumab 1050: Participants received a single dose of capecitabine 1000 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg IV infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
- Capecitabine 1250 + Pertuzumab 1050: Participants received a single dose of capecitabine 1250 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg IV infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Capecitabine 825 Plus (+) Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Started | 5 | 7 | 7
Completed | 2 | 2 | 6
Not Completed | 3 | 5 | 1
Not completed — Insufficient Therapeutic Response | 3 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Refused Treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) Population included all participants who received any amount of the study medication. The baseline analysis population represents participants from all three cohorts.
Groups:
- Capecitabine + Pertuzumab: Participants received a single dose of capecitabine either 825, 1000 or 1250 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg IV infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of the Combination of Pertuzumab and Capecitabine
Description: MTD was defined as the highest tolerated dose combination of capecitabine (825 mg, 1000 mg or 1250 mg) and pertuzumab, without causing Dose Limiting Toxicities (DLTs). DLTs were defined as follows: 1) Any non-hematological toxicity greater than or equal to (≥) Grade 3 according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 except for fever, chills and flu-like symptoms, in spite of adequate toxicity management; 2) Grade 4 neutropenia lasting > 7 days; 3) Febrile neutropenia; 4) Thrombocytopenia Grade 4 or any thrombocytopenia requiring platelet transfusion; 5) Any subjectively intolerable toxicity felt by the investigator to be related to either one of the compounds. Participants who withdrew from the study without completing the first treatment cycle for reasons other than DLT were not considered evaluable for DLT. MTD was measured in mg/m^2.
Time Frame: Cycle 1 (3 Weeks)
Population: The Safety Population included all participants who received any amount of study medication and who had at least one post-baseline safety follow-up.
Measure: Number; unit: mg/m^2
Groups:
- Capecitabine + Pertuzumab: Participants received a single dose of capecitabine either 825,1000 or 1250 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg IV infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
mg/m^2 | 1250

2. Secondary Outcome: Percentage of Participants With DLTs
Description: DLTs were defined as follows: 1)Any non-hematological toxicity greater than or equal to (≥) Grade 3 according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 except for fever, chills and flu-like symptoms, in spite of adequate toxicity management; 2) Grade 4 neutropenia lasting > 7 days; 3) Febrile neutropenia; 4) Thrombocytopenia Grade 4 or any thrombocytopenia requiring platelet transfusion; 5) Any subjectively intolerable toxicity felt by the investigator to be related to either one of the compounds. Participants who withdrew from the study without completing the first treatment cycle for reasons other than DLT were not considered evaluable for DLT.
Time Frame: Cycle 1 (3 Weeks)
Population: Safety population
Measure: Number; unit: percentage of participants
Groups:
- Capecitabine 825 Plus (+) Pertuzumab 1050: Participants received a single dose of capecitabine 825 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg intravenous (IV) infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Arm/Group | Capecitabine 825 Plus (+) Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Number analyzed (Participants) | 5 | 6 | 7
percentage of participants | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Plasma Half-Life (t1/2) of Pertuzumab
Description: The biological half-life or terminal half-life of pertuzumab is the time in days it takes for it to lose half of its pharmacologic activity. t1/2 was measured in days.
Time Frame: Cycle 1: Days 2, 5, 8 and 15 Postdose; Cycle 2: Day 1 at drug administration, predose and 15 minutes postdose, and Predose on Days 8, 15 and 22
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
days | 14.6 (41.0)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Pertuzumab
Description: Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and prior to the administration of a second dose and was measured as nanograms per milliliter (ng/mL).
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
ng/mL | 355111 (59051)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Pertuzumab
Description: Tmax is defined as the time after administration of a drug when the maximum plasma concentration is reached; when the rate of absorption equals the rate of elimination. Tmax was measured in days.
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
days | 0.137 (0.076)

6. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurement (AUC 0-last) of Pertuzumab
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC0-last is calculated from time 0 (prior to administration of medication) to last measured data point. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC was measured as ng*day/mL.
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
ng*day/mL | 2742561 (743598)

7. Secondary Outcome: AUC From Time Zero to Infinity (AUC 0-infinity) of Pertuzumab
Description: The AUC0-infinity is calculated from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC is measured as nanograms times days per milliliter (ng*day/mL).
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
ng*day/mL | 4096501 (1282130)

8. Secondary Outcome: Apparent Volume of Distribution of Pertuzumab
Description: The volume of distribution at steady state (Vss), also known as apparent volume of distribution, is a pharmacological, theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma. Vss was measured in mL
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
mL | 5202 (1007)

9. Secondary Outcome: Apparent Total Clearance of Pertuzumab
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It is measured as milliliters per day (mL/day).
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Capecitabine + Pertuzumab
Number analyzed (Participants) | 18
mL/day | 283.0 (98.0)

10. Secondary Outcome: Plasma Half-Life of Capecitabine and it's Metabolites When Given Alone and in Combination With Pertuzumab
Description: Capecitabine is a novel oral fluoropyrimidine carbamate that is preferentially converted to the cytotoxic moiety fluorouracil (5-fluorouracil; 5-FU) in target tumour tissue through a series of 3 metabolic steps through the intermediate metabolites 5'-deoxy-5-fluorocytidine (5'-DFCR), 5'-deoxy-5-fluorouridine (5'-DFUR), and α-fluoro-β-alanine (FBAL). The biological half-life or terminal half-life is the time in days it takes for it to lose half of its pharmacologic activity.
Time Frame: Day -7: Predose, 30 minutes, 1, 2, 3, 4, 5, 6 and 10 hours postdose; Cycle 1 Day 1: Predose, 0 and 30 minutes, 1, 2, 3, 4, 5, 6 and 10 hours Postdose
Population: ITT population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Capecitabine 825 + Pertuzumab 1050: Participants received a single dose of capecitabine 825 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg intravenous (IV) infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Arm/Group | Capecitabine 825 + Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Number analyzed (Participants) | 5 | 6 | 7
hours
  Capecitabine Alone 5'-DFCR | 0.89 (0.27) | 0.82 (0.28) | 0.82 (0.23)
  Capecitabine Alone 5'-DFUR | 0.75 (0.26) | 0.76 (0.23) | 0.66 (0.09)
  Capecitabine Alone 5-FU | 0.67 (0.22) | 0.64 (0.13) | 0.70 (0.16)
  Capecitabine Alone Capecitabine | 0.54 (0.19) | 0.40 (0.10) | 0.36 (0.11)
  Capecitabine Alone FBAL | 2.54 (0.30) | 2.69 (0.39) | 3.08 (0.78)
  Capecitabine + Pertuzumab 5'-DFCR | 0.78 (0.38) | 0.76 (0.18) | 0.75 (0.14)
  Capecitabine + Pertuzumab 5'-DFUR | 0.62 (0.13) | 0.73 (0.21) | 0.79 (0.28)
  Capecitabine + Pertuzumab 5-FU | 0.73 (0.40) | 0.67 (0.14) | 0.80 (0.35)
  Capecitabine + Pertuzumab Capecitabine | 0.42 (0.14) | 0.62 (0.28) | 0.54 (0.28)
  Capecitabine + Pertuzumab FBAL | 2.59 (0.64) | 2.58 (0.57) | 2.81 (0.44)

11. Secondary Outcome: Maximum Plasma Concentration of Capecitabine and it's Metabolites When Given Alone and in Combination With Pertuzumab
Description: Capecitabine is an oral fluoropyrimidine carbamate that is preferentially converted to the cytotoxic moiety 5-FU in target tumour tissue through a series of 3 metabolic steps through the intermediate metabolites 5'-DFCR, 5'-DFUR, and FBAL. Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and prior to the administration of a second dose and is measures as nanograms per milliliter (ng/mL).
Time Frame: as for outcome 10
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Capecitabine 825 + Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Number analyzed (Participants) | 5 | 6 | 7
ng/mL
  Capecitabine Alone 5'-DFCR | 4508 (2317) | 7687 (1443) | 8647 (3254)
  Capecitabine Alone 5'-DFUR | 5274 (1832) | 7657 (2708) | 10311 (3323)
  Capecitabine Alone 5-FU | 201 (94) | 355 (119) | 369 (107)
  Capecitabine Alone Capecitabine | 4802 (3159) | 9112 (6189) | 7543 (2944)
  Capecitabine Alone FBAL | 3214 (396) | 3963 (947) | 5290 (576)
  Capecitabine + Pertuzumab 5'-DFCR | 4909 (2518) | 3917 (1411) | 6569 (2827)
  Capecitabine + Pertuzumab 5'-DFUR | 5736 (1831) | 4103 (1595) | 8683 (4142)
  Capecitabine + Pertuzumab 5-FU | 219 (106) | 187 (92) | 345 (214)
  Capecitabine + Pertuzumab Capecitabine | 8060 (4800) | 3367 (1741) | 4731 (3198)
  Capecitabine + Pertuzumab FBAL | 3674 (1121) | 3498 (809) | 5136 (843)

12. Secondary Outcome: Time to Maximum Plasma Concentration of Capecitabine and it's Metabolites When Given Alone and in Combination With Pertuzumab
Description: Capecitabine is a novel oral fluoropyrimidine carbamate that is preferentially converted to the cytotoxic moiety fluorouracil (5-fluorouracil; 5-FU) in target tumour tissue through a series of 3 metabolic steps through the intermediate metabolites 5'-deoxy-5-fluorocytidine (5'-DFCR), 5'-deoxy-5-fluorouridine (5'-DFUR), and α-fluoro-β-alanine (FBAL). Tmax is defined as the time after administration of a drug when the maximum plasma concentration is reached; when the rate of absorption equals the rate of elimination.
Time Frame: as for outcome 10
Population: ITT population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Capecitabine 825 + Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Number analyzed (Participants) | 5 | 6 | 7
hours
  Capecitabine Alone 5'-DFCR | 1.3 (0.66) | 0.82 (0.26) | 1.05 (0.51)
  Capecitabine Alone 5'-DFUR | 1.3 (0.66) | 0.76 (0.49) | 1.05 (0.51)
  Capecitabine Alone 5-FU | 1.3 (0.66) | 0.64 (0.49) | 1.05 (0.51)
  Capecitabine Alone Capecitabine | 1.2 (0.75) | 0.4 (0.28) | 0.77 (0.35)
  Capecitabine Alone FBAL | 2.4 (0.55) | 2.69 (0.41) | 2.21 (0.40)
  Capecitabine + Pertuzumab 5'-DFCR | 0.9 (0.65) | 1.42 (0.66) | 1.86 (1.32)
  Capecitabine + Pertuzumab 5'-DFUR | 1.0 (0.61) | 2.0 (1.10) | 1.86 (1.32)
  Capecitabine + Pertuzumab 5-FU | 0.9 (0.65) | 1.84 (1.17) | 1.93 (1.24)
  Capecitabine + Pertuzumab Capecitabine | 0.7 (0.28) | 1.17 (0.40) | 1.15 (0.62)
  Capecitabine + Pertuzumab FBAL | 2.6 (0.90) | 3.16 (1.17) | 2.50 (1.39)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded continuously from Day -7 until 4 weeks after the final visit.
Groups:
- Capecitabine 825 + Pertuzumab 1050: Participants received a single dose of capecitabine 825 mg/m^2 orally on Day -7 and subsequently on Days 1 to 14 of each 3-week cycle administered twice daily. Participants also received pertuzumab on Day 1 of each 3-week cycle as a fixed-dose of 1050-mg IV infusion until progression of the disease, occurrence of unacceptable toxicity or withdrawal of consent.
Arm/Group | Capecitabine 825 + Pertuzumab 1050 | Capecitabine 1000 + Pertuzumab 1050 | Capecitabine 1250 + Pertuzumab 1050
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6 | 1/7
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine 825 + Pertuzumab 1050 (N=5) | Capecitabine 1000 + Pertuzumab 1050 (N=6) | Capecitabine 1250 + Pertuzumab 1050 (N=7)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine 825 + Pertuzumab 1050 (N=5) | Capecitabine 1000 + Pertuzumab 1050 (N=6) | Capecitabine 1250 + Pertuzumab 1050 (N=7)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 7
Nausea (Gastrointestinal disorders) | 4 | 4 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 3 | 4
Mucosal inflammation (General disorders) | 0 | 2 | 4
Pyrexia (General disorders) | 0 | 2 | 2
Oedema Peripheral (General disorders) | 2 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1
Lethargy (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Depressed mood (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 4
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.